CLINICAL TRIAL: NCT06296108
Title: Risk Factors for Acute Kidney Injury in Patients Undergoing Total Joint Arthroplasty
Brief Title: Risk Factors for Acute Kidney Injury in Patients Undergoing Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sanem Cakar Turhan, Associate professor, MD, Ankara University
Other Study IDs: I05-310-22
Record Dates: First submitted 2024-02-26; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Acute Kidney Injury; Arthroplasty
Keywords: arthroplasty; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: acute kidney injury — The incidence of acute kidney injury was determined in patients included to the study

SUMMARY:
The authors aimed to determine the risk factors associated with postoperative acute kidney injury in patients undergoing total joint arthroplasty.

DETAILED DESCRIPTION:
Aim: The primary aim of the current study is to determine the risk factors associated with postoperative acute kidney injury in patients undergoing total joint arthroplasty. Considering that this patient group is mostly composed of advanced age and comorbid patients, the secondary aim of the study is to identify risky patients with predictable risk factors and to chart a way to make preoperative optimizations of the patients before developing postoperative complications.

Materials and Methods: Patients who underwent joint arthroplasty between 2015 and 2020 in Ankara University Faculty of Medicine, Department of Orthopedics and Traumatology were included. Within the scope of the study, patients' gender, age, weight, height, body mass index values, smoking, American Society of Anesthesiologist (ASA) score, Charlson-Comorbidity Index score (CCI), type of operation, duration of surgery, presence of intraoperative hypotension, anesthesia method , diabetes, hypertension, coronary artery disease, presence of congestive heart failure, presence of preoperative anemia, preoperative uric acid and albumin level, use of nephrotoxic agents in the perioperative period, basal creatinine and glomerular filtration rate (GFR) values, platelet suspension in the perioperative period, erythrocyte suspension, Amounts of fresh frozen plasma transfusions, postoperative creatinine at 24 hours - 48 hours - discharge, GFR values and Kidney Disesae Improving Global Outcomes (KDIGO) scores, length of hospital stay and length of stay in the intensive care unit were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 18 years old undergoing arthroplasty surgery

Exclusion Criteria:

* Known acute renal failure or chronic renal failure
* Patients aged below 18 years old
* Patients refusing to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 years old undergoing arthroplasty surgery
Sampling Method: Non-Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury in patients undergoing arthroplasty surgery | Retrospective between 2015-2020
  To determine the incidence of acute kidney injury in patients undergoing arthroplasty surgery

SECONDARY OUTCOMES:
Risk factors causing acute kidney injury in patients undergoing arthroplasty surgery | Retrospective between 2015-2020
  To determine the risk factors causing acute kidney injury in patients undergoing arthroplasty surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sanem Çakar Turhan, Assoc. Prof., Study Chair — Ankara University Medical School, Department of Anesthesiology and ICU; Hazal Nur Tezel Kılıc, Specialist, Principal Investigator — Ankara University Medical School, Department of Anesthesiology and ICU; Suheyla Karadag Erkoc, Assoc. Prof., Principal Investigator — Ankara University Medical School, Department of Anesthesiology and ICU; Hakan Kocaoglu, Assoc. Prof., Principal Investigator — Ankara University Medical School, Department of Orthopedics and Traumatology Surgery
Locations (1):
- Ankara University Medical School Anesthesiology and ICU Department, Ankara, Turkey (Türkiye)